CLINICAL TRIAL: NCT05877404
Title: Practice Patterns Among Gynecologic Oncologists on Tumor Genetic Testing in Endometrial Cancer
Status: Terminated | Type: Observational
Why Stopped: This was a national survey of physicians. Per the protocol, they were only allowed to be contacted twice and they received less surveys back than anticipated.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00097221; WFBCCC 99323 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH); NCI-2023-05554 (Other: CTRP)
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Cancer
Keywords: Genetic testing
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecologic Oncologists: Gynecologic Oncologists and gynecologic oncology fellows-in-training from around the world, who are members of the Society of Gynecologic Oncology (SGO).
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — Survey on practice patterns surrounding tumor genetic testing in endometrial cancer.

SUMMARY:
In order to formulate strategies to improve adherence to best practice guidelines, as well as utilization of novel therapies, investigators must understand current practice patterns surrounding tumor genetic testing in endometrial cancer. The aim is to survey a representative sample of gynecologic oncologists who belong to the society of gynecologic oncology, via an email survey, to better understand current practices surrounding tumor genetic testing as well as determine if there have been any changes to practice since the publication of recent trials on the use of immune-checkpoint inhibitors in endometrial cancer.

DETAILED DESCRIPTION:
Primary Objective: Proportion of physicians reporting the use of different tumor genetic testing strategies among newly diagnosed endometrial cancer patients.

Secondary Objectives:

* Explore the use of informed consent in tumor genetic testing in endometrial cancer
* Explore clinician confidence in utilizing tumor genetic testing to guide treatment decisions.
* Explore the impact of recent publications regarding immunotherapy on the use of tumor genetic testing in endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Society of Gynecologic Oncology
* Gynecologic Oncologist or Gynecologic Oncology Fellow-in-Training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Gynecologic Oncologists and gynecologic oncology fellows-in-training from around the world, who are members of the Society of Gynecologic Oncology (SGO).
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of providers reporting the use of different tumor genetic testing strategies among newly diagnosed endometrial cancer patients | 4 months
  The primary outcome is to estimate the percentage of providers who report the use of different tumor testing strategies. Investigators will calculate the frequencies of responses to each testing strategy and then compare the percentage of physicians who choose different strategies, using a chi-square or Fisher's exact test.

SECONDARY OUTCOMES:
Frequency of providers using different strategies of informed consent in tumor genetic testing in endometrial cancer | 4 months
  Investigators will calculate the number of frequencies of different tumor testing informed consent strategies among physicians.
Number of providers reporting confidence in utilizing tumor genetic testing to guide treatment decisions | 4 months
  Investigators will calculate the number of providers who are very confident, moderately confident, a little confident or not at all confident in their ability to explain tumor testing strategies and results.
Number of providers who change their counseling or testing strategies for endometrial cancer | 4 months
  Investigators will compare the number of providers who have changed their counseling or testing strategy based on their familiarity with recent publications regarding immune-checkpoint inhibitors in advanced and recurrent endometrial cancer using a chi-square or Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, PhD, MPH, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No